CLINICAL TRIAL: NCT06554470
Title: Local Versus Systemic Methotrexate in Management of Uterine Ectopic Pregnancy: A Randomized Trial
Brief Title: Local vs Systemic Methotrexate in Management of Uterine Ectopic Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Nabil Ageez, Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR751/7/24
Record Dates: First submitted 2024-08-11; First posted 2024-08-15 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Local; Systemic; Methotrexate; Uterine Ectopic Pregnancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic Methotrexate (Experimental): Patients will receive systemic methotrexate (intramuscular; 50 mg/m2 body weight).
  Interventions: Drug: Systemic Methotrexate
- Local Methotrexate (Experimental): Patients will receive local methotrexate (25 mg methotrexate as a fixed dose).
  Interventions: Drug: Local Methotrexate

INTERVENTIONS:
Drug: Systemic Methotrexate — Patients will receive systemic methotrexate (intramuscular; 50 mg/m2 body weight).
  Arms: Systemic Methotrexate
Drug: Local Methotrexate — Patients will receive local methotrexate (25 mg methotrexate as a fixed dose).
  Arms: Local Methotrexate

SUMMARY:
This study aims to compare local and systemic methotrexate in the management of uterine ectopic pregnancy regarding the duration of beta human chorionic gonadotropin (hCG) clearance and need for further management options.

DETAILED DESCRIPTION:
Ectopic pregnancy is considered a life-threatening condition which requires immediate intervention. Owing to the advancements in medical technology, ectopic pregnancy can now be diagnosed in the early stages.

Methotrexate (MTX) is an antimetabolite drug showing a competitive reversible binding concerning natural dihydrofolates and acting as an inhibitor of the dihydrofolate-reductase (DHFR), a key enzyme synthesizing the tetrahydrofolates needed for the synthesis of purine and pyrimidine rings.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 40 years.
* Women with uterine ectopic pregnancy (interstitial pregnancy, cervical pregnancy, or cesarean scar pregnancy).
* Gestational age is less than 9 weeks, the embryo size is smaller than 10 mm, and the serum beta-human chorionic gonadotropin (β-hCG) levels are less than 10,000 mIU/mL.

Exclusion Criteria:

* Patients with basal beta hCG levels less than 1500 mIU/Ml.
* Any contraindications to MTX as a hepatic disorder, renal disorder and thrombocytopenia
* Diabetes mellitus.
* Severe vaginal bleeding or hemodynamic changes or hemoperitoneum.
* History of cancer.
* Ascites.
* Pleural effusion.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with uterine ectopic pregnancy
Enrollment: 34 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Time for serum b-hCG remission | Post intervention for 3 months
  Time for serum b-hCG remission will be recorded to be less than 20 iu/ml.

SECONDARY OUTCOMES:
Success rate | Post intervention for 3 months
  Success rate will be recorded.
Time for uterine-mass disappearance | Post intervention for 3 months
  Time for uterine-mass disappearance will be recorded.
Hospitalization time | 15 days after intervention
  Hospitalization time will be recorded from admission till discharge from hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.